CLINICAL TRIAL: NCT05941806
Title: Prophylactic Use of Tamsulosin in the Prevention of Post-operative Urinary Retention in Men After Rectum Resection: a Double-blind Placebo-controlled Clinical Trial
Brief Title: Prophylactic Use of Tamsulosin in the Prevention of Post-operative Urinary Retention in Men After Rectum Resection
Acronym: R-POUR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Fédération des médecins résidents du Québec (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Projet 2023-6826
Record Dates: First submitted 2023-05-12; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Urinary Retention; Colorectal Surgery; Rectal Resection; Post-operative Urinary Retention; Tamsulosin
MeSH Terms: conditions — Urinary Retention | interventions — Tamsulosin; Glucose

STUDY DESIGN:
Intervention Model Description: Our study will be a phase III double-blind randomized clinical trial. A period of 12 to 24 months is planned for recruitment. The primary outcomes are the incidence of postoperative urinary retention in men undergoing rectal resection and the efficacy of prophylactic tamsulosin to prevent this type of complication.
  The secondary outcomes are the length of stay between experimental and placebo groups, the number of urinary catheterizations, the number of urine catheter reinsertions and total duration of urinary catheter being in-situ.
Who Masked: Participant, Care Provider
Masking Description: Patients randomized to the intervention group will receive 0.4 mg tamsulosin capsules, administered orally, once a day for 5 days before surgery, the morning of surgery and the day after surgery. Patients assigned to the placebo group will receive glucose capsules according to the same protocol. The glucose capsules will be manufactured by the pharmacy of the CHU de Quebec
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group receiving Tamsulosin (Active Comparator): Patients randomized to the intervention group will receive 0.4 mg tamsulosin capsules, administered orally, once a day for 5 days before surgery, the morning of surgery and the day after surgery. The steady-state plasma concentration of tamsulosin is reached after 4 to 5 consecutive doses, which justify the administration duration of 5 days preoperatively. The total duration of administration of tamsulosin was established at 7 days since the study of Patel et al. showed a significant reduction in POUR after 7 days of administration.
  Interventions: Drug: pr Sandoz Tamsulosin
- Group receiving Placebo (Placebo Comparator): Patients assigned to the placebo group will receive glucose capsules according to the same protocol. The glucose capsules will be manufactured by the pharmacy of the CHU de Quebec.
  Interventions: Drug: Glucose

INTERVENTIONS:
Drug: pr Sandoz Tamsulosin — Sandoz Tamsulosin, the study drug, is an alpha1-adrenergic blocking agent approved by Health Canada for men with bladder outlet obstruction symptoms associated with benign prostatic hyperplasia.
  Other Names: Tamsulosin hydrochloride
  Arms: Group receiving Tamsulosin
Drug: Glucose — Patients assigned to the placebo group will receive glucose capsules according to the same protocol. The glucose capsules will be manufactured by the pharmacy of the CHU de Quebec
  Arms: Group receiving Placebo

SUMMARY:
The study will be a phase III double-blind randomized clinical trial. Participants will be recruited from the Department of General Surgery of the CHU de Québec - Saint-François-d'Assise and Hôtel-Dieu de Québec. The primary outcomes are the incidence of postoperative urinary retention in men undergoing rectal resection and the efficacy of prophylactic tamsulosin to prevent this type of complication.The secondary outcomes are the length of stay between experimental and placebo groups, the number of urinary catheterizations, the number of urine catheter reinsertions and total duration of urinary catheter being in-situ.

DETAILED DESCRIPTION:
Participants will be recruited consecutively during their preoperative visit to the outpatient clinic. Participants will be followed by a logbook throughout the follow-up period, as well as by their surgical and research teams. Follow-up will begin on the first day of pre-operative medication and will end 30 days after surgery. Patients randomized to the intervention group will receive 0.4 mg tamsulosin capsules, administered orally, once a day for 5 days before surgery, the morning of surgery and the day after surgery. Patients assigned to the placebo group will receive glucose capsules according to the same protocol. The glucose capsules will be manufactured by the pharmacy of the CHU de Quebec. All patients will have a foley catheter inserted for surgery. Their urinary catheter (foley catheter) will be removed at 6:00 AM the day after their surgery (post-operative day 1). The diagnosis of urinary retention will be suspected by a member of the patient's medical team if a patient has no miction for 8 hours or more or 4 hours or more after removal of foley catheter or after the surgery. In these cases, a portable bladder scanner will be used. The diagnosis of post-operative urinary retention (POUR) will be confirmed in two situations: 1. If there is 500ml of urine or more in the bladder 2. If there is 300ml or urine or more with at least 1 of the following symptoms: urge to urinate with inability to urinate, suprapubic pain or signs and symptoms of delirium. When the diagnosis of POUR will be made, urine will be removed from the bladder using an in/out bladder catheterization. After using a bladder catheterization, a portable bladder scanner will be used again if a patient has no spontaneous urination for the first 4 hours after catheterization. A second bladder catheterization will be done once again in the same two situations as described above. At the third bladder catheterization, a urinary (foley) catheter will be inserted. The catheter will be left in place for 24h before attempting a trial of void. A member of the medical team will then collect the information in the patient's logbook and medical record. Adherence to drug intake will be self-reported to the patient's diary. The patient can indicate why he missed one or more doses of the drug. Patients will receive a list of potential side effects of tamsulosin with their logbook. The side effects will be self-reported by the patient to the logbook each day. The patients' logbook will be analysed by the research team. Two independent reviewers of the research team will collect the other variables. They will perform a standardized retrospective revision of the medical records according to a pre-established data collection grid. We will perform an intention-to-treat analysis in this prospective randomized study. Postoperative urinary retention remains a frequent complication and causes significant discomfort in men undergoing rectal resection. The decrease in its incidence could then significantly reduce the number of bladder catheterizations required postoperatively, and thus reduce the incidence of complications associated with it. The prevention of POUR will allow patients a more harmonious postoperative recovery, limited in inconvenience and side effects, and an earlier return home. Ultimately, the health care costs associated with this postoperative complication may be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* 18 years and older
* Scheduled for rectal resection during the study period.

Exclusion Criteria:

* Patients undergoing revisional surgery
* Patients taking alpha-blocker medication,
* Patients who have an indwelling urinary catheter,
* Patients who have undergone urinary tract surgery,
* Patients who will have an intraoperative trauma of the urinary tract,
* Patients who will keep their urinary catheter for more than 24 hours after surgery,
* Patients who have an intolerance to alpha-blocking drugs or who take one of the following drugs (potential interaction): anti-retroviral, antifungal, clarithromycin, erythromycin, paroxetine, terbinafine, cimetidine, coumadin or phosphodiesterase inhibitors.
* Patients who will have an epidural anesthesia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative urinary retention | During the length of hospital stay: up to two weeks
  Incidence of postoperative urinary retention in men undergoing rectal resection

SECONDARY OUTCOMES:
Length of stay | During hospital stay: up to two weeks
  Length of stay between experimental and placebo groups
Number of urinary catheterizations | During hospital stay: up to two weeks
  Number of bladder catheterization
Number of urine catheter reinsertions | During hospital stay: up to two weeks
  Number of urine catheter reinsertions
Total duration of urinary catheter being in-situ | During hospital stay: up to two weeks
  Number of days a foley catheter will be in place

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Beauchamp, MD, Principal Investigator
Locations (2):
- Canada (2):
  - Hotel Dieu de Quebec, Québec, Quebec
  - Hôpital Saint-François d'Assise, Québec

IPD SHARING:
Plan to Share IPD: No